CLINICAL TRIAL: NCT02213341
Title: Impact of Vaccination on Th2 Immunity in Infancy
Status: Terminated | Type: Observational
Why Stopped: Lack of enrollment.
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Consortium of Food Allergy Research (Other)
Responsible Party: Sponsor
Other Study IDs: DAIT CoFAR9
Record Dates: First submitted 2014-08-07; First posted 2014-08-11 (Estimated); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Food Hypersensitivity
Keywords: Milk Allergy; Egg Allergy; Peanut Allergy; Infant Vaccination
MeSH Terms: conditions — Food Hypersensitivity; Milk Hypersensitivity; Egg Hypersensitivity; Peanut Hypersensitivity | interventions — Blood Specimen Collection; Phlebotomy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Positive blood test to milk, egg, and/or peanut: Family history to atopy
  Interventions: Procedure: Skin prick allergen test; Procedure: Blood draw
- Negative blood test to allergy: A negative skin prick test to egg, milk, and peanut and a negative Immunoglobulin E (IgE) to egg, milk, and peanut.
  Interventions: Procedure: Skin prick allergen test; Procedure: Blood draw

INTERVENTIONS:
Procedure: Skin prick allergen test — To test for hypersensitivity to milk, egg, or peanut
Procedure: Blood draw
  Other Names: venipuncture

SUMMARY:
The purpose of this study is to assess the responses in the immune system of infants after they receive the vaccine against diphtheria, tetanus, and pertussis (DTaP). The investigators will do this by studying the immune cells and allergy responses in the blood prior to and after receipt of the third DTaP vaccine.

DETAILED DESCRIPTION:
This is a single-site study of infants who are scheduled to receive their third series (~6 month) vaccinations, as routine care, to investigate whether the diphtheria, tetanus, and pertussis (DTaP) vaccination has an effect on specific immunoglobulin E (IgE) levels to milk, egg, or peanut. Infants will be assigned to one of two groups depending on the infant's sensitization to milk, egg, and peanut.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent from parent/guardian
* General good health without other known need for blood draws that would conflict with the study volume requirements
* Aged 5 months - 7 months, any race/ethnicity, any gender
* Subjects must not have yet received their third DTaP vaccination, which typically is given at 6 months of age. Subjects must have previously received two doses of the DTaP vaccination, at ages 2 months and 4 months
* Willingness to return for follow-up testing as defined in the protocol and consent if screening tests indicate eligibility
* Group 1 participants must have all of the following:

  * A negative skin prick test to egg, milk, and peanut
  * A negative IgE to egg, milk, and peanut
* Group 2 participants must have all of the following:

  * A positive family history of allergic disease
  * Atopic Dermatitis not requiring prescription medication
  * A positive IgE to milk, egg, and/or peanut

If Group 1 enrollment is completed first, participants must have all of the following to be enrolled in Group 2:

* A family history of atopy
* Atopic dermatitis not requiring prescription medication

If Group 2 enrollment is completed first, participants must have all of the following to be enrolled in Group 1:

-No personal or family history of atopic disease

Exclusion Criteria:

* History of anemia requiring any treatment
* Previous allergic reaction to any food, defined as itching, rash, hives, swelling, vomiting, diarrhea, sneezing, rhinorrhea, wheezing, breathing difficulty, or passing out immediately after food ingestion.
* Evidence of non-IgE-mediated reaction to milk or soy (i.e. milk/soy protein intolerance) or evidence of food protein induced enterocolitis syndrome (FPIES)
* Severe atopic dermatitis (liberally defined as requiring prescription medication)
* Unable to obtain serum sample for determination of egg, milk and peanut IgE levels
* Use of short-acting anti-histamines (diphenhydramine, etc.) more than one time within 3 days of skin testing or on the day of skin testing
* Any history of intravenous or oral steroid medication
* Known underlying immune defect/deficiency or bleeding disorder

Ages: 5 Months to 7 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Infants who are scheduled to receive their ~6 month (third dose of primary series) vaccines including the DTaP vaccine as part of routine care.
Sampling Method: Probability Sample
Enrollment: 77 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2016-06-14 (Actual); Study Completion 2016-06-14 (Actual)

PRIMARY OUTCOMES:
Allergen-specific IgE | baseline and day 28
  Magnitude of increase of allergen-specific IgE. For each child, the maximum allergen-specific IgE change to milk, egg, or peanut will be considered as the primary endpoint.

CONTACTS AND LOCATIONS:
Overall Officials: Hugh A. Sampson, MD, Principal Investigator — Icahn School of Medicine at Mt. Sinai; Scott Sicherer, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

REFERENCES:
- See also: National Institute of Allergy and Infectious Diseases (NIAID) — https://www.niaid.nih.gov/
- See also: Division of Allergy, Immunology, and Transplantation (DAIT) — https://www.niaid.nih.gov/about/dait
- See also: Consortium of Food Allergy Research (CoFAR) — http://www.cofargroup.org/